CLINICAL TRIAL: NCT06581562
Title: Open-label Single-Center Study to Evaluate the Safety and Efficacy of Combining Rituximab and AB-101 in B-cell Associated Autoimmune Diseases.
Acronym: IRIS-RD-01
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: IRIS Research and Development, LLC (Other)
Collaborators: Artiva Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRIS-RD-01
Record Dates: First submitted 2024-08-02; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Rheumatoid Arthritis; Pemphigus Vulgaris; Granulomatosis With Polyangiitis; Systemic Lupus Erythematosus
MeSH Terms: conditions — Arthritis, Rheumatoid; Pemphigus; Granulomatosis with Polyangiitis; Lupus Erythematosus, Systemic | interventions — Rituximab; Cyclophosphamide; fludarabine

STUDY DESIGN:
Intervention Model Description: Open-label Single-Center Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): Arm 1 - Subjects with Rheumatoid Arthritis
  Interventions: Drug: AB-101; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Fludarabine
- Arm 2 (Experimental): Arm 2- Pemphigus Vulgaris
  Interventions: Drug: AB-101; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Fludarabine
- Arm 3 (Experimental): Arm 3 - Systemic Lupus Erythematosus
  Interventions: Drug: AB-101; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Fludarabine
- Arm 4 (Experimental): Arm 4- Subjects with Granulomatosis with polyangiitis / microscopic polyangiitis
  Interventions: Drug: AB-101; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: AB-101 — Subjects in all 4 indications will receive only one cycle of treatment.
  Subjects with RA, PV or SLE will receive one cycle of treatment as follows:
  1. Fludarabine: 25 mg/m2 on Day 1, Day 2 and Day 3.
  2. Cyclophosphamide: 1000 mg/m2 on Day 3
  3. Rituximab: 1000 mg on Day 1 and Day 15
  4. AB-101: 1B NK cells (AlloNK) on Day 6, Day 13 and Day 20
  Subjects with GPA and MPA will receive one cycle of treatment as follows:
  1. Fludarabine: 25 mg/m2 on Day 1, Day 2, and Day 3.
  2. Cyclophosphamide: 1000 mg/m2 on Day 3
  3. Rituximab: 375 mg/m2 on Day -2, Day 6, Day 13, and Day 20
  4. AB-101: 1B NK cells (AlloNK) on Day 6, Day 13, and Day 20 The first dose of AB-101 should be administered at least 48 hours after the last infusion of the lymphodepletion regimen.
  Other Names: ALLONK; RITUXIMAB; CYCLOPHOSPHAMIDE; FLUDARABINE
Drug: Rituximab — Subjects in all 4 indications will receive only one cycle of treatment.
  Subjects with RA, PV or SLE will receive one cycle of treatment as follows:
  1. Fludarabine: 25 mg/m2 on Day 1, Day 2 and Day 3.
  2. Cyclophosphamide: 1000 mg/m2 on Day 3
  3. Rituximab: 1000 mg on Day 1 and Day 15
  4. AB-101: 1B NK cells (AlloNK) on Day 6, Day 13 and Day 20
  Subjects with GPA and MPA will receive one cycle of treatment as follows:
  1. Fludarabine: 25 mg/m2 on Day 1, Day 2, and Day 3.
  2. Cyclophosphamide: 1000 mg/m2 on Day 3
  3. Rituximab: 375 mg/m2 on Day -2, Day 6, Day 13, and Day 20
  4. AB-101: 1B NK cells (AlloNK) on Day 6, Day 13, and Day 20 The first dose of AB-101 should be administered at least 48 hours after the last infusion of the lymphodepletion regimen.
Drug: Cyclophosphamide — Subjects in all 4 indications will receive only one cycle of treatment.
  Subjects with RA, PV or SLE will receive one cycle of treatment as follows:
  1. Fludarabine: 25 mg/m2 on Day 1, Day 2 and Day 3.
  2. Cyclophosphamide: 1000 mg/m2 on Day 3
  3. Rituximab: 1000 mg on Day 1 and Day 15
  4. AB-101: 1B NK cells (AlloNK) on Day 6, Day 13 and Day 20
  Subjects with GPA and MPA will receive one cycle of treatment as follows:
  1. Fludarabine: 25 mg/m2 on Day 1, Day 2, and Day 3.
  2. Cyclophosphamide: 1000 mg/m2 on Day 3
  3. Rituximab: 375 mg/m2 on Day -2, Day 6, Day 13, and Day 20
  4. AB-101: 1B NK cells (AlloNK) on Day 6, Day 13, and Day 20 The first dose of AB-101 should be administered at least 48 hours after the last infusion of the lymphodepletion regimen.
Drug: Fludarabine — Subjects in all 4 indications will receive only one cycle of treatment.
  Subjects with RA, PV or SLE will receive one cycle of treatment as follows:
  1. Fludarabine: 25 mg/m2 on Day 1, Day 2 and Day 3.
  2. Cyclophosphamide: 1000 mg/m2 on Day 3
  3. Rituximab: 1000 mg on Day 1 and Day 15
  4. AB-101: 1B NK cells (AlloNK) on Day 6, Day 13 and Day 20
  Subjects with GPA and MPA will receive one cycle of treatment as follows:
  1. Fludarabine: 25 mg/m2 on Day 1, Day 2, and Day 3.
  2. Cyclophosphamide: 1000 mg/m2 on Day 3
  3. Rituximab: 375 mg/m2 on Day -2, Day 6, Day 13, and Day 20
  4. AB-101: 1B NK cells (AlloNK) on Day 6, Day 13, and Day 20 The first dose of AB-101 should be administered at least 48 hours after the last infusion of the lymphodepletion regimen.

SUMMARY:
This study will evaluate the safety and activity of AB-101 in combination with rituximab in B-cell associated autoimmune diseases where rituximab is currently FDA approved (e.g., Rheumatoid Arthritis (RA), Pemphigus Vulgaris (PV), Granulomatosis with polyangiitis (GPA)/microscopic polyangiitis (MPA) as a therapeutic, or is recommended (e.g., in Systemic Lupus Erythematosus (SLE) as a cornerstone for disease management.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria (applicable to subjects in all 4 studied indications)

1. Males or female subjects, ≥ 18 years of age at the time of signing informed consent.
2. Ability to understand the requirements of the study.
3. Willingness to provide written informed consent.
4. Willingness to comply with the study protocol procedures.
5. Women of childbearing potential and all male participants must agree to use two acceptable methods of contraception together to avoid pregnancy. The following are examples of acceptable methods of contraception including:

   1. Established use of oral, inserted, injected, or implanted hormonal methods of contraception.
   2. Correctly placed copper containing intrauterine device (IUD).
   3. Male condom or female condom used WITH a spermicide (i.e., foam, gel, film, cream, suppository).
   4. Male sterilization with appropriately confirmed absence of sperm in the post-vasectomy ejaculate.
   5. Bilateral tubal ligation or bilateral salpingectomy.
6. Oral steroids will be tapered to <20 mg/day of prednisone (or equivalent) at least 1 week prior to the first study treatment. The tapering schedule will be at the discretion of the Investigator.
7. Subjects must have a predicted diffusing capacity for carbon monoxide (DLCO) of >60% and a forced expiratory volume 1 (FEV1) >70% at screening.
8. Left ventricular ejection fraction (LVEF) ≥ 45% by Echocardiogram. Rituximab and AB-101 in autoimmune diseases Clinical Study Protocol V. 1.1 Confidential Page 11 of 101 April 16, 2024
9. Baseline laboratory values fulfilling the following requirements to demonstrate adequate hematologic, renal, and hepatic function:

RA PV MPA / GPA SLE Absolute neutrophil count (/mm3)

* 1500
* 1500
* 1500
* 1500 Platelets (/mm3)
* 100,000
* 100,000
* 100,000
* 75,000 Hemoglobin (g/dL)
* 9
* 9
* 9
* 8 Creatinine clearance (mL/min/1.73 m2)
* 60
* 60
* 60
* 60 Total serum bilirubin (mg/dL) < 2.5 < 2.5 < 2.5 < 2.5 Liver transaminases (AST/ALT/ALP)

  ≤ 3x ULN

  ≤ 3x ULN
  * 3x ULN
  * 3x ULN Additional Disease-specific Inclusion Criteria Rheumatoid Arthritis

    1. Documented diagnosis of RA, meeting the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria for RA (Kay, 2012).

    2. Have had prior treatment for a period of at least 12 weeks with a biologic disease-modifying anti-rheumatic drugs (bDMARD e.g., infliximab, rituximab, etanercept, tocilizumab)) and/or a targeted synthetic disease-modifying anti-rheumatic drugs (tsDMARD e.g., baricitinib, tofacitinib)) and were deemed refractory by either:
    1. In the opinion of the Investigator, there was a lack of benefit to at least two bDMARDs or one bDMARD and one tsDMARDs. Lack of benefit may include inadequate improvement in joint counts, physical function, or disease activity.
    2. Intolerance to at least two lines of prior therapy, including bDMARDs and/or tsDMARDs.

       3. Minimum of 6 swollen joint counts (SJC) and 6 tender joint counts (TJC). Pemphigus Vulgaris
       1. Confirmed diagnosis of pemphigus vulgaris with active lesions.
       2. Positive for anti-desmoglein Dsg1 or Dsg3.
       3. Pemphigus Disease Area Index score of > 10%.
       4. Subjects will have tried and failed at least 12 weeks of treatment of immunosuppressive or biologic standard-of-care agent (methotrexate, azathioprine, mycophenolate mofetil (MMF) or mycophenolic acid (MPA) and corticosteroids, and/or 12 weeks of therapy with IV Gamma globulin treatments with an exposure of 12 weeks to be considered resistant/refractory and will be included in this study.

          Granulomatosis with polyangiitis (GPA) / microscopic polyangiitis (MPA)

       <!-- -->

       1. Clinical diagnosis of granulomatosis with polyangiitis (GPA) or microscopic polyangiitis (MPA).
       2. Presence of cytoplasmic Antineutrophil cytoplasmic antibody (c-ANCA) or proteinase-3 (PR3-ANCA) or myeloperoxidase ANCA (MPO-ANCA)
       3. Have ≥ 1 "major" item, or ≥ 3 "other" items, or ≥ 2 renal items on the Birmingham Vasculitis Activity Score Version 3 (BVASv3).
       4. For GPA/MPA, subjects will have tried and failed at least 12 weeks of treatment of immunosuppressive (Cyclophosphamide, mycophenolate mofetil (MMF) or mycophenolic acid (MPA) and corticosteroids), or a biologic standard-of-care agent such as Rituximab will be included in this study.

       Systemic Lupus Erythematous
       1. Diagnosis of SLE according to the 2019 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) Classification Criteria.
       2. Total systemic lupus erythematosus disease activity index (SLEDAI-2K) ≥ 8 at screening excluding alopecia, mucosal ulcers, and fever.
       3. Positive for anti-double-stranded deoxyribonucleic acid (dsDNA) antibodies.
       4. For SLE, subjects will have tried and failed at least 12 weeks of 2 conventional therapies which, at the discretion of the investigator, includes antimalarials, corticosteroids, immunosuppressive agents, such as mycophenolate mofetil, Methotrexate, Azathioprine, as well as biologic agents such as Belimumab, Anifrolumab, and Rituximab.

       The following criteria for standard-of-care therapies must be met:

    <!-- -->

    1. If receiving antimalarial drugs (e.g., hydroxychloroquine, chloroquine, quinacrine), must have used the medication for ≥ 12 weeks prior to first study treatment and at a stable dose for a minimum of 6 weeks prior to first administration of AB-101.
    2. If receiving immunomodulatory drugs (mycophenolate mofetil [MMF]/mycophenolic acid ≤ 2 g/day, azathioprine/6 mercaptopurine (AZA/6 MP) ≤ 2 mg/kg/day, leflunomide ≤ 40 mg/day, methotrexate (MTX) ≤ 25 mg/wk with concomitant folic acid [recommend ≥ 5 mg/wk]), calcineurin inhibitor, and/or cyclosporin A, receiving a stable dose for at least 12 weeks prior to the first administration of AB-101.

       Oral corticosteroid (OCS) <20 mg/day prednisone or equivalent started at least 12 weeks prior to first study treatment and at a stable dose for at least 4 weeks prior to first administration of study treatment. It must be planned that the background standard-of-care treatment remains at a stable dose throughout the Screening Period.

       Exclusion Criteria:

       General Exclusion Criteria (applicable to subjects in all 4 studied indications) 1. Subjects who received Cyclophosphamide within 3 months 2. Laboratory values outside the protocol-defined range at screening, unless the PI documents that the abnormal laboratory value does not compromise patient safety or interfere with the study's goals.

       3. Known hypersensitivity or contraindication to any drug products or any component of the drug products they plan to receive (e.g., cyclophosphamide, fludarabine, rituximab, AB-101).

       4. History of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies or DMSO (Dimethyl sulfoxide).

       5. Prior treatment with any B-cell targeted therapy within 3 months of the start of the planned lymphodepletion regimen (e.g., rituximab or other anti-CD20, anti-CD19, anti-CD22 monoclonal antibodies) 6. Prior treatment with any autologous or allogeneic cell therapy approach using genetically modified immune cells (e.g., T, NK, macrophages, or gamma-delta T cells modified with chimeric antigen receptors (CAR)).

       7. Received any of the following within 6 months of the start of the planned lymphodepletion regimen:

    <!-- -->

    1. Immunoglobulin replacement therapies (IV or SC)
    2. Plasmapheresis. 8. History of a major organ transplant (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplant, or are due to receive such transplantation.

       9. Known past or current malignancy except for cervical carcinoma of stage 1B or less, noninvasive basal cell or squamous cell skin carcinoma, Noninvasive, superficial bladder cancer, Prostate cancer with a current prostate specific antigen (PSA) level < 0.1 ng/m, Any curable cancer with a complete response duration of > 2 years 10. Any history of a B cell malignancy, even if subjects have achieved a complete response.

       11. Known clinically significant cardiac disease: Within the prior 6 months of signing the informed consent form, onset of unstable angina pectoris or acute myocardial infarction; congestive heart failure (grade III or IV as classified by the New York Heart Association), pericarditis present during screening or at baseline, heart rate-corrected QT interval (QTcF) prolongation > 470 msec at screening, unless secondary to stable conduction disorders (e.g., left bundle-branch block) 12. Unresolved toxicities from prior therapy, defined as having not resolved to Grade ≤ 1, or to the levels dictated in the eligibility criteria.

       13. Have clinical evidence of significant unstable or uncontrolled acute or chronic diseases not due to RA, PV, GPA/MPA, SLE (e.g., cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, renal, neurological, malignancy, or infectious diseases) which, in the opinion of the principal investigator, could confound the results of the study or put the subject at undue risk.

       14. Have a planned surgical procedure or a history of any other medical disease (e.g., cardiopulmonary), laboratory abnormality, or condition (e.g., poor venous access) that, in the opinion of the principal investigator, makes the subject unsuitable for the study.

       15. Have any signs or symptoms of illness/infection or have received any vaccinations (live or inactivated) within 6 weeks of Day 1.

       16. Have current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within ≤ 1 year prior to Day 1.

       17. Human immunodeficiency virus (HIV) infection, based on laboratory testing performed during the screening period.

       18. Currently pregnant or lactating (breast feeding must not be started within 6 months of the last dose of AB-101).

       19. Any other considerations that might interfere with the assessment of safety or efficacy, or that the investigator deems inappropriate for inclusion.

       20. Any medical, psychological, familial, or sociological condition that, in the Investigator's opinion, would impair the subject's ability to receive study treatment or comply with study requirements.

       21. Severe disease progression or health deterioration within 2 weeks of Day 1 that, in the opinion of the Investigator, could impair the ability of the subject to receive study treatment or comply with study requirements.

       22. Known past or current clinically significant lung disease. 23. History of, or current, chronic pulmonary disease (e.g., COPD, asthma, etc.) not meeting DLCO and FEV1 eligibility criteria 24. Pulmonary manifestations of underlying autoimmune disease that may compromise pulmonary function.

       25. History of tobacco exposure of ≥ 5 pack years 26. Subjects with a prior history of hypogammaglobulinemia or with low IgG levels (< 600 mg/dL). Subjects who have received Intravenous Immunoglobulins (IVIG) for any reason in the 3 months prior to screening will be excluded.

       27. Current use of tobacco product Additional Disease specific Exclusion Criteria Rheumatoid Arthritis
       1. History of a rheumatologic autoimmune disease other than RA (except secondary Sjögren's)
       2. Significant systemic involvement secondary to RA (e.g., vasculitis, pulmonary fibrosis, Felty's syndrome)
       3. Other arthritis, including Juvenile idiopathic arthritis (JIA) or idiopathic arthritis diagnosed before the age of 16 years; Psoriatic Arthritis; Axial spondylarthritis or any other disease associated with inflammatory arthritis; Active fibromyalgia with pain symptoms or signs that would interfere with clinical assessments for RA.

       Pemphigus Vulgaris
       1. Any condition, including potential flares or new infected or non-infected lesions that would, in the investigator's judgment, interfere with full participation in the study.

       Granulomatosis with polyangiitis (GPA) / microscopic polyangiitis (MPA) 1. Any other multi-system autoimmune disease. 2. Have required significant ongoing management of infections Systemic Lupus Erythematous
       1. Drug-induced lupus.
       2. Participants with a history of severe anti-phospholipid syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events and relationship to study drug | From the time of consent through 104 weeks after initiation of study treatment
  We will evaluate the Incidence of adverse events and relationship to study drug
Incidence of Serious Adverse Events (SAE) and causality assessment | From the time of consent through 104 weeks after initiation of study treatment
  We will evaluate the Incidence of adverse events and relationship to study drug
Total hospitalizations, duration of hospitalizations through the course of the study | From the time of consent through 104 weeks after initiation of study treatment
  We will evaluate the Incidence of adverse events and relationship to study drug

SECONDARY OUTCOMES:
RA: Change From Baseline in DAS28 at Week 12 and 24 | Week 12 through 24
  RA: Change From Baseline in DAS28 at Week 12 and 24
PV: Change from baseline in the Pemphigus Disease Area Index (PDAI) at Week 12 and 24 | Week 12 through 24
  PV: Change from baseline in the Pemphigus Disease Area Index (PDAI) at Week 12 and 24
GPA / MPA: Change from baseline in the Birmingham Vasculitis Activity Score at Week 12 and 24 | Week 12 through 24
  GPA / MPA: Change from baseline in the Birmingham Vasculitis Activity Score at Week 12
SLE: Change from baseline in the SLE Disease Activity Index (SLEDAI) at Week 12 and 24 | Week 12 through 24
  SLE: Change from baseline in the SLE Disease Activity Index (SLEDAI) at Week 12 and 24

OTHER OUTCOMES:
Pharmacokinetics and Immunogenicity | at baseline and according to the scheduled of assessments
  Blood samples for pharmacokinetic analysis and immunogenicity will be collected according to the SoA
Patient Reported Outcomes | from the time of consent through 104 weeks after initiation of styudy treatment
  Patient Reported Outcomes
Pharmacodynamic Biomarkers | from the time of consent through 104 weeks after initiation of styudy treatment
  The following biomarkers will be measured at baseline and according to the scheduled of assessments. Autoantibodies: ANA, anti-dsDNA, aCL (IgG, IgM, IgA isotypes), anti-Sm, and anti- C1q 2. Serum immunoglobulin isotypes: IgA, IgG, IgM 3. Serum complement (C3, C4) 4. Serum cytokines/chemokines, urinary biomarkers 5. Peripheral B cell subsets, T and NK lymphocytes 6. DSG 1 and DSG 3 autoantibodies

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo J. Valenzuela, M.D., Principal Investigator — IRIS Research and Development, LLC; Kathy I. Perez, M.D., Study Director — IRIS Research and Development, LLC
Locations (1):
- IRIS Research and Development, LLC, Plantation, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided